CLINICAL TRIAL: NCT06594458
Title: To Reduce the Separation of the Mother-newborn Dyad in the First Day of Life Through the Implementation of a New Procedure in the Delivery Room
Brief Title: New Procedure to Reduce Mother-newborn Separation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6113
Record Dates: First submitted 2023-10-23; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-10

CONDITIONS: Neonatal Disease
MeSH Terms: conditions — Infant, Newborn, Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neonatal Respiratory Distress Arm (Experimental): Newborn manifesting tachypnea or respiratory distress in the delivery room (that responds to supplementary oxygen with FiO2 <30% and without the need for mechanical ventilation) are placed in a preheated incubator with the required oxygen concentration (if necessary) and carefully monitored by medical and nursing clinicians.
  Interventions: Procedure: Observation of newborn with respiratory distress in the delivery room

INTERVENTIONS:
Procedure: Observation of newborn with respiratory distress in the delivery room — Newborn manifesting tachypnea or respiratory distress at birth (that responds to supplementary oxygen with FiO2 <30% and without the need for mechanical ventilation) are placed in a preheated incubator with the required oxygen concentration (if necessary) and carefully monitored by medical and nursing clinicians. A clinical evaluation will be carried out every 15 minutes, with the detection of vital parameters. In case of clinical improvement and suspension of oxygen therapy, the newborn will be transferred to the Neonatal Observation Ward to perform multiparameter monitoring of vital signs up to 6 hours of life and then be reunited with the mother. In case of clinical worsening, a bedside thoracic ultrasound will be carried out and depending on the result and the lung ultrasonography score, it will be evaluated whether to continue the observation in the delivery room or to admit the newborn in the Neonatal Care, Neonatal Sub-Intensive Care or Neonatal Intensive care Units

SUMMARY:
The goal of this single-centre interventional study without medication neither device (for procedure) is to limit the separation between mother and newborn by implementing a new procedure for the management of the newborn with respiratory distress in the delivery room.

The main questions it aims to answer are:

* Is it possible to reduce Neonatal Intensive Care Unit admissions within 24 hours of life by applying this new procedure, thus limiting separation between mother and newborn?
* Does the implementation of this procedure, reducing mother-newborn separation, improves the rate of exclusive breastfeeding?

Newborns with respiratory distress at birth will be evaluated in the delivery room in a dedicated pre-heated incubator, providing additional oxygen if necessary. In case of improvement they will be reunited with the mother, in case of worsening a thoracic ultrasound will be performed to assess the severity and possible hospitalization in Neonatal Intensive Care Unit

DETAILED DESCRIPTION:
This procedure provides that newborn infants, who at 15 minutes of life manifest tachypnea or respiratory distress (that responds to supplementary oxygen with FiO2 <30% and without the need for mechanical ventilation) they are placed in a preheated incubator with the required oxygen concentration (if necessary) and carefully monitored by medical and nursing clinicians. A clinical evaluation will be carried out every 15 minutes, with the detection of vital parameters, such as heart rate, oxygen saturation and respiratory rate. In case of clinical improvement and suspension of oxygen therapy, the newborn will be transferred to the Neonatal Observation Ward to perform multiparameter monitoring of vital signs up to 6 hours of life and then be reunited with the mother. In case of clinical worsening, a bedside thoracic ultrasound will be carried out and depending on the result and the Lung Ultrasonography score, it will be evaluated whether to continue the observation in the delivery room or hospitalize the newborn in the Neonatal Care, Neonatal Sub-Intensive Care or Neonatal Intensive care Units.

ELIGIBILITY:
Inclusion Criteria:

* Infants born by elective cesarean section, with gestational age ≥34 weeks, weight at birth ≥2000 grams, manifesting mild respiratory distress with need for oxygen at FiO2 ≤30%
* Signature by both parents of an informed consent

Exclusion Criteria:

* Multiple pregnancy
* Need for invasive respiratory assistance
* Need for resuscitation at birth
* Criteria for perinatal asphyxiation
* Fetal pathology
* Failure by both parents to sign up for informed consent

Ages: 1 Minute to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 142 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Limit the separation between mother and newborn | 3 hours
  Newborn manifesting respiratory distress at birth are placed in a preheated incubator with the required oxygen concentration (if necessary). A clinical evaluation will be carried out every 15 minutes, with the detection of vital parameters. In case of clinical improvement and suspension of oxygen therapy, the newborn will be transferred to the Neonatal Observation Ward to perform multiparameter monitoring of vital signs up to 6 hours of life and then be reunited with the mother. In case of clinical worsening, a bedside thoracic ultrasound will be carried out it will be evaluated whether to continue the observation in the delivery room or to admit the newborn in the Neonatal Care or Neonatal Intensive care Units

SECONDARY OUTCOMES:
Exclusive Breastfeeding rate | 3 days
  To evaluate improvement in exclusive breastfeeding as a result of the new procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Agostino Gemelli IRCCS, UOC Neonatologia, Roma, Italy